CLINICAL TRIAL: NCT03831230
Title: Constitution of ex Vivo Ovarian Tumor Models for the Validation of the Interest of Innovative Therapies and the Search for Tumor or Circulating Biomarkers Predictive of Treatment Response
Acronym: OVAREX
Status: Completed | Type: Observational
Sponsor: Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-A02152-53
Record Dates: First submitted 2019-01-28; First posted 2019-02-05 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Ovarian Cancer
Keywords: ex vivo; predictive tests; tumor models
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Urination; Tumor Burden

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Genetic: collection of blood, urine, tumor and ascite samples — collection of blood, urine, tumor and ascite samples during ovarian surgery

SUMMARY:
Development of ex vivo models of ovarian cancer, fallopian tubes or peritoneum.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old.
* Patient with ovarian cancer, carcinoma of the fallopian tubes, or histologically proven peritoneum. All FIGO stages are accepted for the study.
* Patient to be managed by surgery (laparoscopy and / or laparotomy).

Exclusion Criteria:

* Pregnant woman
* Persons deprived of liberty or guardianship (including curatorship)
* History of any other clinically active malignancy in the last 5 years prior to inclusion

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patient with ovarian cancer, carcinoma of the fallopian tubes, or histologically proven peritoneum. All FIGO stages are accepted for the study.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2019-03-07 (Actual); Primary Completion 2025-02-27 (Actual); Study Completion 2025-02-27 (Actual)

PRIMARY OUTCOMES:
Rates of exploitable ex vivo tumor, blood and urine samples for performing predictive tests | Collection of blood, urine, tumor and ascite samples at the time of ovarian surgery
  Number and quality of tumor, blood and urine samples that can be used to perform predictive tests of the response to treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Centre François BACLESSE, Caen, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Thorel L, Divoux J, Lequesne J, Babin G, Morice PM, Florent R, Desmartin G, Lecouflet L, Marde Alagama C, Leconte A, Clarisse B, Briand M, Rouzier R, Gaichies L, Martin-Francoise S, Le Brun JF, Denoyelle C, Vigneron N, Jeanne C, Blanc-Fournier C, Leman R, Vaur D, Figeac M, Meryet-Figuiere M, Joly F, Weiswald LB, Poulain L, Dolivet E. The OVAREX study: Establishment of ex vivo ovarian cancer models to validate innovative therapies and to identify predictive biomarkers. BMC Cancer. 2024 Jun 7;24(1):701. doi: 10.1186/s12885-024-12429-w. PMID 38849726